CLINICAL TRIAL: NCT00850642
Title: The Efficacy of Orally Administered GSK2190915 as an add-on to Current Therapy in Subjects With Moderate to Severe Asthma Who Have Elevated Sputum Neutrophils
Brief Title: GSK2190915 Moderate to Severe Asthma Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112046; 2008-007244-33 (EudraCT Number)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Sputum cell counts; Neutrophils; Severe Asthma; ICS; Inhaled corticosteroids
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 12 day repeat dosing with placebo
  Interventions: Drug: Placebo
- GSK2190915 100mg (Experimental): 12 day repeat dosing treatment phase with 100mg GSK2190915.
  Interventions: Drug: GSK2190195 100mg

INTERVENTIONS:
Drug: GSK2190195 100mg — GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor.
  Arms: GSK2190915 100mg
Drug: Placebo — Placebo :
  2% (w/w) Ethanol, sucralose (5 mg/100 mL of oral solution) to 100 % (w/w) aqueous sodium carbonate buffer (0.010 M, pH 9-10)
  Arms: Placebo

SUMMARY:
A randomised, double-blind, placebo-controlled, parallel group study to evaluate the effect of treatment with GSK2190915, a FLAP inhibitor, as add-on to current inhaled corticosteroid therapy in patients with moderate to severe asthma with elevated sputum neutrophils.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Males and females aged 18 to 65 years inclusive.
* Body mass index within the range 18.5-37.0 kilograms/metre2 (kg/m2).
* An established clinical history of Asthma in accordance with the definition by the GINA Guidelines [GINA, 2006]. Subjects should have at screening or within the last year documented reversibility (>12 %) to short acting bronchodilator, or positive methacholine challenge, or positive histamine challenge (PC20 <8mg/ml).
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with documented (medical report verification) hysterectomy or double oophrectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy; childbearing potential and agrees to use one of the contracception methods listed in Section 8.1 for an appropriate period of time prior to the start of dosing and until 3 months after last dose.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 3 months after the last dose.
* Subject with moderate to severe asthma with forced expiratory volume in one second (FEV1) ≥ 50% of predicted.
* Subject who are on regular inhaled corticosteroids without or in combination with a regular long acting Beta 2 Agonist. The dose should be stable for at least 4 weeks before screening.
* Subjects who are taking a minimum of FP 250mg BID or equivalent.
* Persistent sputum neutrophilia defined by sputum neutrophils ≥ 65% with TTC < 15 million cells/g with no evidence of eosinophilia (sputum eosinophils < 2%). Persistent is defined as the criteria being met at screening (or within the 6 months preceding screening) and on visit 1.
* Signed and dated written informed consent is obtained from the subject
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Past or present disease, which as judged by the investigator or medical monitor, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, gastrointestinal disease, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (excluding asthma but including but not confined to chronic bronchitis, emphysema, bronchiectasis, eosinophilic bronchitis or pulmonary fibrosis).
* Clinically significant abnormalities in safety laboratory analysis at screening.
* Subject has uncontrolled hypertension or is hypertensive at screening. Hypertension at screening is defined as persistent systolic BP >150 mmHg or diastolic BP > 90mmHg.
* History of asthma exacerbations or acute intercurrent respiratory illness (viral respiratory syndrome, bronchitis, pneumonia) for a four week period before the screening visit
* History of life-threatening asthma, defined as an asthma episode that required intubations and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* Subject is unable to abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-histamines and anti-asthma, anti-rhinitis or hay fever medication, with the exception of ICS, LABA and short action beta agonists, from 14 days before screening until the follow-up visit unless in the opinion of the Investigator and sponsor the medication will not interfere with the study
* Administration of oral or injectable steroids within 6 weeks of screening.
* The subject has participated in a study with a new molecular entity during the previous 3 months or has participated in 4 or more clinical studies in the previous 12 months prior to the first dosing day.
* Administration of anti -leukotrienne therapies for 14 days before screening and during the study.
* Administration of any vaccinations within 1 month of screening or during the study.
* Administration of biological therapies within 3 months of the screening visit or during the study
* Subject is undergoing allergen desensitisation therapy.
* Administration of OATP1B1 substrates from 2 weeks before dosing, and until all follow-up assessments are completed.
* There is a risk of non-compliance with study procedures.
* History of blood donation (500 mL) within 3 months of starting the clinical study.
* The subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female. One unit of alcohol is defined as a medium (125 ml) glass of wine, half a pint (250 ml) of beer or one measure (25 ml) of spirits.
* The subject has a screening QTc value of >450msec, PR interval outside the range 120 to 220msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave).
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV antibodies.
* The subject has a positive pre-study urine drug or urine or breath alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbituates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06-26 (Actual); Primary Completion 2010-06-02 (Actual); Study Completion 2010-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Canada (4):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- United Kingdom (4):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated prior to completion due to difficulties in recruiting the required participants. A total of 7 asthmatic participants completed the study prior to termination. The study was, conducted from 26 June 2009 to 02 June 2010, at three centers in Canada and three centers in the United Kingdom.
Groups:
- Placebo: The eligible participants in this arm were administered with matching placebo, orally, once daily for 12-days.
- GSK2190915: The eligible participants in this arm received GSK2190915 as 100 milligram (mg), orally once daily for 12-days.
Period: Overall Study
Arm/Group | Placebo | GSK2190915
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The eligible participants in this arm were administered with matching placebo, orally once daily for 12-days.
- GSK2190915: The eligible participants in this arm received GSK2190915 as 100 mg, orally, once daily for 12-days.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2190915 | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (12.12) | 57.8 (6.65) | 55.3 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Numbers of Neutrophils in Induced Sputum-Absolute Neutrophil Count
Description: The neutrophils play an important role in participants with more severe asthma. The reduction in number of neutrophils in induced sputum was evaluated to study the effect of treatment with repeat oral doses of GSK2190915, in asthma participants. Sputum samples were evaluated at central laboratory. The samples were rejected, if the weight was less than 100 grams (g), or if excessive cell degeneration or due to excessive squamous cells and insufficient inflammatory cells. The total cell count of neutrophil was reported as total cell count × 10^6 /g.
Time Frame: Day -9 to -7, Day 1, Day 12 and follow-up (Day 24-28)
Population: All Subject Population was defined as all participants who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Giga cells per g
Groups:
- GSK2190915: The eligible participants in this arm received GSK2190915 as 100 mg, orally once daily for 12-days
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Giga cells per g
  Day -9 to -7 | 5.205 (2.8415) | 3.096 (2.6093)
  Day 1: number analyzed (Participants) | 2 | 3
  Day 1 | 3.142 (3.2449) | 14.667 (20.8291)
  Day 12: number analyzed (Participants) | 2 | 3
  Day 12 | 13.534 (13.6394) | 0.396 (0.0801)
  Follow-up: number analyzed (Participants) | 2 | 3
  Follow-up | 5.359 (1.1681) | 2.995 (3.6389)

2. Primary Outcome: Percentage of Neutrophils in Induced Sputum
Description: The neutrophils play an important role in participants with more severe asthma. The reduction in number of neutrophils in induced sputum was evaluated to study the effect of treatment with repeat oral doses of GSK2190915, in asthma participants. Sputum samples were evaluated at central laboratory. The samples were rejected, if the weight was less than 100 g, or if excessive cell degeneration or due to excessive squamous cells and insufficient inflammatory cells. The total cell count of neutrophil was reported as percentage of cells.
Time Frame: Day -9 to -7, Day 1, Day 12 and follow-up (Day 24-28)
Population: All Subject Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Percentage of neutrophils
  Day -9 to -7 | 84.00 (9.469) | 74.88 (2.269)
  Day 1, pre-dose: number analyzed (Participants) | 2 | 3
  Day 1, pre-dose | 68.00 (10.607) | 74.77 (18.351)
  Day 12, 2 hour: number analyzed (Participants) | 2 | 3
  Day 12, 2 hour | 86.30 (16.263) | 56.33 (19.732)
  Follow-up: number analyzed (Participants) | 2 | 3
  Follow-up | 65.75 (0.071) | 78.33 (14.640)

3. Secondary Outcome: Assessment of FEV1 on Visit 2, 3 and Visit 4
Description: FEV1 is the amount of air which can be forcefully exhaled in 1 second. It was assessed using a spirometry. Due to early termination of the study, the data of individual participants is reported.
Time Frame: Visit 2 (Day 1), visit 3 (Day 5 to 7) and visit 4 (Day 12)
Population: All Subject population. Individual participant data reported, due to early termination of study. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Measure: Number; unit: Liters
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Liters
  Particpant 1, Day 1, Pre-dose: number analyzed (Participants) | 1 | 0
  Particpant 1, Day 1, Pre-dose | 2.33 |
  Particpant 1, Day 1, 2 hour: number analyzed (Participants) | 1 | 0
  Particpant 1, Day 1, 2 hour | 2.55 |
  Participant 1, Day 5 to 7/ Visit 3: number analyzed (Participants) | 1 | 0
  Participant 1, Day 5 to 7/ Visit 3 | 2.56 |
  Participant 1, Day 12, Pre-dose: number analyzed (Participants) | 1 | 0
  Participant 1, Day 12, Pre-dose | 2.83 |
  Particpant 1, Day 12, 2 hour: number analyzed (Participants) | 1 | 0
  Particpant 1, Day 12, 2 hour | 2.77 |
  Particpant 2, Day 1, Pre-dose: number analyzed (Participants) | 1 | 0
  Particpant 2, Day 1, Pre-dose | 2.88 |
  Particpant 2, Day 1, 2 hour: number analyzed (Participants) | 1 | 0
  Particpant 2, Day 1, 2 hour | 3.06 |
  Participant 2, Day 5 to 7/Visit 3: number analyzed (Participants) | 1 | 0
  Participant 2, Day 5 to 7/Visit 3 | 2.96 |
  Participant 2, Day 12, Pre-dose: number analyzed (Participants) | 1 | 0
  Participant 2, Day 12, Pre-dose | 3.26 |
  Particpant 2, Day 12, 2 hour: number analyzed (Participants) | 1 | 0
  Particpant 2, Day 12, 2 hour | 3.14 |
  Particpant 3, Day 1, Pre-dose: number analyzed (Participants) | 1 | 0
  Particpant 3, Day 1, Pre-dose | 1.65 |
  Particpant 3, Day 1, 2 hour: number analyzed (Participants) | 1 | 0
  Particpant 3, Day 1, 2 hour | 1.98 |
  Participant 3, Day 5 to 7/ Visit 3: number analyzed (Participants) | 1 | 0
  Participant 3, Day 5 to 7/ Visit 3 | 1.92 |
  Participant 3, Day 12, Pre-dose: number analyzed (Participants) | 1 | 0
  Participant 3, Day 12, Pre-dose | 1.81 |
  Particpant 3, Day 12, 2 hour: number analyzed (Participants) | 1 | 0
  Particpant 3, Day 12, 2 hour | 1.83 |
  Particpant 4, Day 1, Pre-dose: number analyzed (Participants) | 0 | 1
  Particpant 4, Day 1, Pre-dose |  | 1.97
  Particpant 4, Day 1, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 4, Day 1, 2 hour |  | 2.14
  Participant 4, Day 5 to 7/ Visit 3: number analyzed (Participants) | 0 | 1
  Participant 4, Day 5 to 7/ Visit 3 |  | 2.22
  Participant 4, Day 12, Pre-dose: number analyzed (Participants) | 0 | 1
  Participant 4, Day 12, Pre-dose |  | 2.02
  Particpant 4, Day 12, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 4, Day 12, 2 hour |  | 1.90
  Particpant 5, Day 1, Pre-dose: number analyzed (Participants) | 0 | 1
  Particpant 5, Day 1, Pre-dose |  | 2.24
  Particpant 5, Day 1, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 5, Day 1, 2 hour |  | 2.78
  Participant 5, Day 5 to 7/ Visit 3: number analyzed (Participants) | 0 | 1
  Participant 5, Day 5 to 7/ Visit 3 |  | 2.07
  Participant 5, Day 12, Pre-dose: number analyzed (Participants) | 0 | 1
  Participant 5, Day 12, Pre-dose |  | 1.89
  Particpant 5, Day 12, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 5, Day 12, 2 hour |  | 2.02
  Particpant 6, Day 1, Pre-dose: number analyzed (Participants) | 0 | 1
  Particpant 6, Day 1, Pre-dose |  | 1.10
  Particpant 6, Day 1, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 6, Day 1, 2 hour |  | 1.22
  Participant 6, Day 5 to 7/ Visit 3: number analyzed (Participants) | 0 | 1
  Participant 6, Day 5 to 7/ Visit 3 |  | 1.22
  Participant 6, Day 12, Pre-dose: number analyzed (Participants) | 0 | 1
  Participant 6, Day 12, Pre-dose |  | 1.10
  Particpant 6, Day 12, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 6, Day 12, 2 hour |  | 1.19
  Particpant 7, Day 1, Pre-dose: number analyzed (Participants) | 0 | 1
  Particpant 7, Day 1, Pre-dose |  | 1.03
  Particpant 7, Day 1, 2 hour: number analyzed (Participants) | 0 | 1
  Particpant 7, Day 1, 2 hour |  | 1.13
  Participant 7, Day 5 to 7/ Visit 3: number analyzed (Participants) | 0 | 1
  Participant 7, Day 5 to 7/ Visit 3 |  | 1.14
  Participant 7, Day 12, Pre-dose: number analyzed (Participants) | 0 | 1
  Participant 7, Day 12, Pre-dose |  | 1.11

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, or is an important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or a drug-induced liver injury.
Time Frame: From visit 1 (Day -7 to Day -9) to upto follow-up (upto Day 28)
Population: All Subject Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Participants
  Any AE | 2 | 3
  Any SAE | 0 | 0

5. Secondary Outcome: Number of Participants With Vital Sign of Potential Clinical Concern (PCC)
Description: The vital sign measurement included measurement of systolic and diastolic blood pressure alongwith pulse rate. The PCC values reported for systolic blood pressure were < 85 millimeter of mercury (mmHg) and >160 mmHg; that for diastolic was <45 mmHg and >100 mmHg. The PCC values for pulse rate were <40 and > 110 beats per minute. The number of participants with values outside the PCC for systolic, diastolic blood pressure and vitals during the treatment duration were reported.
Time Frame: Visit 2 (Day 1) to Upto follow-up (Day 28)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Participants
  Systolic blood pressure | 0 | 0
  Diastolic blood pressure | 0 | 0
  Heart rate | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: The number of participants with abnormal ECG values were reported. The data was reported as Abnormal clinically significant (CS), abnormal not clinically significant (NCS), and No result.
Time Frame: Visit 2 (Day 1) to Upto follow-up (Day 28)
Population: All Subject Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Participants
  Abnormal NCS, Day 1, pre-dose | 1 | 1
  No results, Day 1 pre-dose 2 | 1 | 0
  No results, Day 1 pre-dose 3 | 1 | 0
  Abnormal NCS, Day 1, pre-dose 2 hour | 1 | 0

7. Secondary Outcome: Number of Participants With Clinical Chemistry Values of PCC
Description: The clinical chemistry parameters evaluated were albumin, calcium, creatinine, glucose, magnesium, phosphorus, potassium, sodium, urea, gamma glutamyl transferase, and bicarbonate. The number of participants with values outside the PCC values were reported. The PCC value observed for bicarbonate was reported.
Time Frame: Visit 2 (Day 1) to Upto follow-up (Day 28)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With Hematology Values of PCC
Description: The hematology parameters evaluated were white blood cells, neutrophils, hemoglobin, hematocrit, platelets and lymphocytes. The number of participants with values outside the PCC values were reported. The PCC value observed for lymphocyte was reported.
Time Frame: Visit 2 (Day 1) to Upto follow-up (Day 28)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: The eligible participants in this arm were administered with matching placebo, once daily for 12-days.
- GSK2190915: The eligible participants in this arm received 100 mg GSK2190915, once daily for 12-days.
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Participants | 0 | 1

9. Secondary Outcome: Plasma Concentration of GSK2190915
Description: The blood samples for analysis of pharmacokinetic parameters were collected at pre-dose and 2 hours post dose on Day 1 and pre-dose trough and 2 hour post dose on Day 12, to evaluate the concentration of the drug GSK2190915 in plasma.
Time Frame: At Day 1, pre-dose; Day 1, 2 hour; Day 12, pre-dose; and Day 12, 2 hour
Population: All Subject Population.
Measure: Mean (Standard Deviation); unit: Nanogram per millilitre
Arm/Group | GSK2190915
Number analyzed (Participants) | 4
Nanogram per millilitre
  Day 1, pre-dose | 0.000 (NA) — For 0.000 dispersion could not be calculated.
  Day 1, 2 hour | 1609.303 (958.4609)
  Day 12, pre-dose | 1073.623 (627.7852)
  Day 12, 2 hour | 2334.238 (1252.5057)

10. Secondary Outcome: Percentage Change From Baseline Urine LTE4 Biomarker
Description: The urine spot samples were collected from the participants at pre-dose on day 1 and trough day 12 for evaluation of LTE4 biomarker. This evaluated the level of inflammation in the airways of the asthma participants. The percentage change from baseline was calculated by dividing the post randomization change by the baseline value from the individual and multiplying by a 100. If either the baseline or post-randomization value is missing, the change from baseline is set to missing. Baseline was defined as Day 1(pre-dose).
Time Frame: Day 1 and Day 12
Population: All subject population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Percent change | 26.22 (89.173) | -89.62 (4.996)

11. Secondary Outcome: Percentage Change From Baseline of LTB4 Biomarker in Plasma
Description: The plasma samples were evaluated for presence of LTB4 biomarkers. The percentage change from baseline was calculated by dividing the post-randomization change by the baseline value from the individual and multiplying by a 100. If either the baseline or post-randomization value is missing, the change from baseline is set to missing. Baseline was defined as Day 1(pre-dose).
Time Frame: Day 1 and Day 12
Population: All subject population.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Percentage change
  Day 1, 2 hour | -24.72 (53.130) | -95.24 (6.711)
  Day 12, pre-dose: number analyzed (Participants) | 3 | 3
  Day 12, pre-dose | 282.81 (452.763) | -95.29 (7.326)
  Day 12, 2 hour: number analyzed (Participants) | 3 | 3
  Day 12, 2 hour | -22.05 (58.391) | -99.23 (1.010)

12. Secondary Outcome: Concentration of LTB4 in Sputum
Description: The concentration of LTB4 levels in sputum were evaluated. However due to early termination of the study, the data was not collected.
Time Frame: Day 1 and Day 12
Population: All Subject Population. Data not collected.
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Concentration of Interleukin (IL)-17 and High-sensitivity C-reactive Protein (hsCRP) in Blood
Description: The blood samples were collected to evaluate the concentration of IL-17 and hsCRP in blood. However due to early termination of the study, the data was not collected.
Time Frame: Day 1 and Day 12
Population: All Subject Population. Data not summarized for this parameter.
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Assessment of Established Markers of Anti-inflammatory Activity in Sputum: the Measurements Will Include IL-17, Neutrophil Elastase, Myeloperoxidase and IL-8
Description: During the study conduct it was observed that the levels of IL-17, measured in both blood and sputum were below limit of quantification; for neutrophil elastase, in sputum no inference could be made as most levels were above the limit of quantification. Thus due to limited amount of data the analysis was not summarized.
Time Frame: Day 1 and Day 12
Population: All Subjects Population. Collected data were below the limit of quantification, so data could not be summarized
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Asthma Control Questionnaire (ACQ) Assessment
Description: ACQ measures the adequacy of asthma control. It includes 5 questions about symptoms of asthma, 1 question about the rescue medication used and 1 about lung function (FEV1% predicted). This is a 7-item scale where the items are equally weighted and the ACQ score is the mean of 7 items which ranges from 0 to 6. 0= Well controlled and 6=extremely poorly controlled. Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma. Thus for ACQ a higher score indicates severe disease and a low score indicative of less severe disease.
Time Frame: At Day 1, Day 5 to 7 and Day 12
Population: All Subject Population.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | GSK2190915
Number analyzed (Participants) | 3 | 4
Scores on scale
  Day 1 | 1.19 (0.218) | 1.57 (0.857)
  Day 5 to 7 | 1.29 (0.286) | 1.50 (0.474)
  Day 12 | 1.14 (0.429) | 1.54 (0.811)

ADVERSE EVENTS:
Time Frame: From visit 1 (Day -7) to upto follow-up (upto Day 28)
Description: All subject population was used to record the AEs.
Arm/Group | Placebo | GSK2190915
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | GSK2190915 (N=4)
Headache (Nervous system disorders) | 1 | 2
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Bacterial test positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulties in recruiting the required participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.